CLINICAL TRIAL: NCT00952367
Title: Prevalence of Nasopharyngeal Carriage of Streptococcus Pneumoniae in Healthy Children Aged 12-18 Months in Six Cities of China
Brief Title: Prevalence of Nasopharyngeal Carriage of Streptococcus Pneumoniae in Healthy Children of 12-18 Months in 6 Cities, China
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-4602
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Streptococcus Pneumoniae Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Per-protocol population: In all, 3641 participants were enrolled; however, 38 were excluded because of violation of inclusion/exclusion criteria and 3 participants were excluded for unavailability of nasopharyngeal swab sample. The record presents demographic and result data for 3600 participants in the per-protocol population. These participants completed collection of the nasopharyngeal swab sample, the Epidemiology questionnaire, and 24 hours safety observation.
  Interventions: Other: Nasopharyngeal swab

INTERVENTIONS:
Other: Nasopharyngeal swab — Nasopharyngeal swab

SUMMARY:
This study is to observe the carriage rate of Streptococcus pneumoniae (S.p.), Haemophilus influenzae Type B (Hib) and Moraxella catarrhalis (M.Cat.) in healthy Chinese children aged 12-18 months in order to estimate the prevalence of pathogens that commonly cause infection in Chinese young children. The antibiotic resistance of all isolates and the serotypes distribution of S.p. isolates will also be tested. Potential risk factors for nasopharyngeal carriage will be collected.

ELIGIBILITY:
Inclusion Criteria

* Healthy children aged 12-18 months

Exclusion Criteria

* Use of antibiotics up to 15 days prior to study inclusion
* Malformation or injury of the nasopharynx that makes the procedure of taking a nasopharyngeal swab impossible
* Children with chronic infectious (chronic otitis media or chronic sinusitis prior to study inclusion.
* Received any pneumococcal vaccine in the past.
* Children who have already provided a NP sample in the same study period.
* Any relevant hemorrhagic disorder.
* Any febrile process (fever ≥ 38°C) at time of screening.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Children 12 to 18 months old
Sampling Method: Non-Probability Sample
Enrollment: 3641 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- China (6):
  - Pfizer Investigational Site, Beijing, Beijing Municipality
  - Pfizer Investigational Site, Dongguan, Guangdong
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Jinan, Shandong
  - Pfizer Investigational Site, Shanghai, Shanghai Municipality

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X1-4602&StudyName=Prevalence%20of%20Nasopharyngeal%20Carriage%20of%20Streptococcus%20Pneumoniae%20in%20Healthy%20Children%20of%2012-18%20Months%20in%206%20Cities%2C%20China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In all, 3641 participants were enrolled; however, 38 were excluded because of violation of inclusion/exclusion criteria and 3 participants were excluded for unavailability of nasopharyngeal swab sample. The record presents demographic and result data for 3600 participants in the per-protocol population.
Groups:
- All Enrolled Participants: Enrolled participants signed the informed consent form, satisfied all screening criteria, and were eligible to enter the study.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 3641
Completed | 3635
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Noncoordination | 1
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 3600
Age Continuous [Mean (Standard Deviation); unit: months] | 14.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1718
  Male | 1882

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Nasopharyngeal Carriage of Streptococcus Pneumoniae
Description: A nasopharyngeal swab sample approached via the nasal route was collected. Swab samples were inoculated directly on plates and transferred to local laboratory for culture and isolation of Streptococcus pneumoniae. Percentage of participants in whom Streptococcus pneumoniae was isolated is reported by site.
Time Frame: Day 1
Population: Per-protocol (PP): Participants who completed collection of nasopharyngeal swab sample, Epidemiology Questionnaire, and 24 hours safety observation. n=number of participants analyzed at that site.
Measure: Number; unit: percentage of participants
Groups:
- Per-protocol Population: Enrolled participants completed collection of the nasopharyngeal swab sample, the Epidemiology questionnaire, and 24 hours safety observation.
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 3600
percentage of participants
  Beijing (n=600) | 12.5
  Shanghai (n=614) | 7.2
  Jinan (n=594) | 16.6
  Nanjing (n=598) | 9.3
  Wuhan (n=596) | 10.5
  Dongguan (n=598) | 18.9

2. Primary Outcome: Percentage of Participants With Serotypes of Streptococcus Pneumoniae
Description: Categories are the serotypes of Streptococcus pneumoniae. NO6A/NO6B belongs to Group 6 but is neither 6A nor 6B. NO23F belongs to Group 23 but is not 23F. NO19A/NO19F belongs to Group 19 but is neither 19A nor 19F. Serotypes G, H, D, I, E, F are results of latex agglutination test, and do not refer to a specific serotype; they cannot be further serotyped by the Quellung reaction. NO(Without capsule) includes all Streptococcus pneumoniae isolates that cannot be serotyped because of no capsule.
Time Frame: Day 1
Population: PP. Number of participants analyzed = number of participants with carriage of Streptococcus pneumoniae isolates.
Measure: Number; unit: percentage of participants
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 451
percentage of participants
  19F | 28.4
  14 | 7.5
  19A | 6.7
  15 | 6.7
  6B | 6.4
  NO6A/NO6B | 3.5
  17 | 2.0
  NO23F | 2.0
  18 | 1.6
  10 | 1.1
  8 | 0.9
  11 | 0.9
  20 | 0.7
  22 | 0.7
  33 | 0.4
  7 | 0.2
  4 | 0.2
  9 | 0.2
  NO19A/NO19F | 0.2
  G | 8.9
  H | 3.1
  D | 0.9
  I | 0.7
  E | 0.7
  F | 0.2
  NO(Without capsule) | 3.5
  23F | 6.0
  6A | 5.8

3. Secondary Outcome: Percentage of Participants With Nasopharyngeal Carriage of Haemophilus Influenzae Type B
Description: A nasopharyngeal swab sample approached via the nasal route was collected. Swab samples were inoculated directly on plates and transferred to local laboratory for culture and isolation of Haemophilus influenzae type B. Percentage of participants in whom Haemophilus influenzae type B was isolated is reported by site.
Time Frame: Day 1
Population: PP. n=number of participants analyzed at that site.
Measure: Number; unit: percentage of participants
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 3600
percentage of participants
  Beijing (n=600) | 4.3
  Shanghai (n=614) | 8.0
  Jinan (n=594) | 5.7
  Nanjing (n=598) | 2.3
  Wuhan (n=596) | 3.4
  Dongguan (n=598) | 4.2

4. Secondary Outcome: Percentage of Participants With Nasopharyngeal Carriage of Moraxella Catarrhalis
Description: A nasopharyngeal swab sample approached via the nasal route was collected. Swab samples were inoculated directly on plates and transferred to local laboratory for culture and isolation of Moraxella catarrhalis. Percentage of participants in whom Moraxella catarrhalis was isolated is reported by site.
Time Frame: Day 1
Population: PP. n=number of participants analyzed at that site.
Measure: Number; unit: percentage of participants
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 3600
percentage of participants
  Beijing (n=600) | 11.7
  Shanghai (n=614) | 11.1
  Jinan (n=594) | 9.8
  Nanjing (n=598) | 7.9
  Wuhan (n=596) | 8.2
  Dongguan (n=598) | 17.4

5. Secondary Outcome: Percentage of Streptococcus Pneumoniae Isolates Resistant to Antibiotics
Description: Categories are types of antibiotics. Penicillin (Old Criteria): Criteria of non-meningitis Streptococcus pneumoniae isolates resistant to penicillin were changed in Clinical Laboratory and Standards Institute (CLSI) in 2008. Criteria in CLSI before 2008 were the old criteria.
Time Frame: Day 1
Population: PP. Number of participants analyzed = number of participants with carriage of Streptococcus pneumoniae.
Measure: Number; unit: percentage of isolates
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 451
percentage of isolates
  Penicillin (Old Criteria) | 18.6
  Penicillin | 1.1
  Amoxicillin/clavulanic acid | 1.1
  Cefuroxime | 23.5
  Cefatriaxone | 4.0
  Azithromycin | 83.6
  Erythromycin | 83.6
  Levofloxacin | 0.2
  Moxifloxacin | 0.0

6. Secondary Outcome: Percentage of Haemophilus Influenzae Type B Isolates Resistant to Antibiotics
Description: Categories are types of antibiotics.
Time Frame: Day 1
Population: PP. Number of participants analyzed = number of participants with carriage of Haemophilus influenzae type B.
Measure: Number; unit: percentage of isolates
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 168
percentage of isolates
  Cefuroxime | 0.0
  Cefatriaxone | 0.0
  Azithromycin | 1.2
  Levofloxacin | 0.0
  Moxifloxacin | 2.4
  Ampicillin | 19.6

7. Secondary Outcome: Percentage of Moraxella Catarrhalis Isolates Resistant to Antibiotics
Description: Categories are types of antibiotics.
Time Frame: Day 1
Population: PP. Number of participants analyzed = number of participants with carriage of Moraxella catarrhalis.
Measure: Number; unit: percentage of isolates
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 396
percentage of isolates
  Cefuroxime | 0.0
  Cefatriaxone | 0.0
  Azithromycin | 21.0
  Levofloxacin | 0.0
  Erythromycin | 22.7

8. Secondary Outcome: Risk Factors Associated With Nasopharyngeal Carriage for Streptococcus Pneumoniae
Description: Risk factors include age of mother bearing (less than or equal to [<=] 30 years versus [vs] more than [>] 30 years); household register (local vs nonlocal); mother's education level (illiteracy, elementary school, junior middle school, senior/vocational high school or technical, college/university vs postgraduate and above); family monthly income per capita (below 600 Chinese Renminbi [RMB], 600 RMB to 1999 RMB, 2000 RMB to 4999 RMB, 5000 RMB to 7999 RMB, 8000 RMB to 9999 RMB vs more than or equal to [>=] 10000 RMB); whether have brothers or sisters (yes vs no).
Time Frame: Day 1
Population: PP
Measure: Mean (Standard Error); unit: relative risk
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 3600
relative risk
  Age of mother bearing, <=30 years vs >30 years | 0.248 (0.070)
  Household register, local vs nonlocal | -0.116 (0.062)
  Mother's education, illiteracy vs postgraduate | 1.087 (0.396)
  Mother's education, elementary vs postgraduate | 0.326 (0.199)
  Mother's education, junior middle vs postgraduate | 0.209 (0.149)
  Mother's education, senior high vs postgraduate | -0.068 (0.157)
  Mother's education, college vs postgraduate | -0.643 (0.175)
  Monthly income, <600 RMB vs >=10000 RMB | 0.508 (0.251)
  Monthly income, 600 to 1999 RMB vs >= 10000 RMB | 0.448 (0.175)
  Monthly income, 2000 to 4999 RMB vs >= 10000 RMB | 0.396 (0.172)
  Monthly income, 5000-7999 RMB vs >= 10000 RMB | -0.230 (0.254)
  Monthly income, 8000 to 9999 RMB vs >= 10000 RMB | -0.834 (0.615)
  Whether have brothers or sisters, no vs yes | -0.331 (0.065)
Statistical Analysis 1: Comparison: Per-protocol Population; Age of mother bearing, <=30 years vs >30 years; Test type: Superiority or Other; p < 0.001, Chi-squared; Degrees of freedom=1, Wald Chi-Square=12.514; Odds Ratio (OR) = 1.641, 95% CI 2-sided [1.247 to 2.159]
Statistical Analysis 2: Comparison: Per-protocol Population; Household register, local vs nonlocal; Test type: Superiority or Other; p = 0.060, Chi-squared; Degrees of freedom=1, Wald Chi-Square=3.529; Odds Ratio (OR) = 0.793, 95% CI 2-sided [0.622 to 1.010]
Statistical Analysis 3: Comparison: Per-protocol Population; Mother's education level, illiteracy vs postgraduate or above; Test type: Superiority or Other; p = 0.006, Chi-squared; Degrees of freedom=1, Wald Chi-Square=7.524; Odds Ratio (OR) = 7.369, 95% CI 2-sided [1.672 to 32.479]
Statistical Analysis 4: Comparison: Per-protocol Population; Mother's education level, elementary school vs postgraduate or above; Test type: Superiority or Other; p = 0.102, Chi-squared; Degrees of freedom=1, Wald Chi-Square=2.671; Odds Ratio (OR) = 3.443, 95% CI 2-sided [1.001 to 11.843]
Statistical Analysis 5: Comparison: Per-protocol Population; Mother's education level, junior middle school vs postgraduate or above; Test type: Superiority or Other; p = 0.159, Chi-squared; Degrees of freedom=1, Wald Chi-Square=1.984; Odds Ratio (OR) = 3.064, 95% CI 2-sided [0.933 to 10.067]
Statistical Analysis 6: Comparison: Per-protocol Population; Mother's education level, senior high school/vocational high school/technical secondary school vs postgraduate or above; Test type: Superiority or Other; p = 0.662, Chi-squared; Degrees of freedom=1, Wald Chi-Square=0.191; Odds Ratio (OR) = 2.321, 95% CI 2-sided [0.710 to 7.589]
Statistical Analysis 7: Comparison: Per-protocol Population; Mother's education level, college/university vs postgraduate or above; Test type: Superiority or Other; p < 0.001, Chi-squared; Degrees of freedom=1, Wald Chi-Square=13.525; Odds Ratio (OR) = 1.306, 95% CI 2-sided [0.399 to 4.277]
Statistical Analysis 8: Comparison: Per-protocol Population; Family monthly income per capita, <=600 RMB vs >=10000 RMB; Test type: Superiority or Other; p = 0.043, Chi-squared; Degrees of freedom=1, Wald Chi-Square=4.095; Odds Ratio (OR) = 2.217, 95% CI 2-sided [0.719 to 6.831]
Statistical Analysis 9: Comparison: Per-protocol Population; Family monthly income per capita, 600 to 1999 RMB vs >=10000 RMB; Test type: Superiority or Other; p = 0.010, Chi-squared; Degrees of freedom=1, Wald Chi-Square=6.549; Odds Ratio (OR) = 2.089, 95% CI 2-sided [0.739 to 5.906]
Statistical Analysis 10: Comparison: Per-protocol Population; Family monthly income per capita, 2000 to 4999 RMB vs >=10000 RMB; Test type: Superiority or Other; p = 0.021, Chi-squared; Degrees of freedom=1, Wald Chi-Square=5.313; Odds Ratio (OR) = 1.983, 95% CI 2-sided [0.704 to 5.583]
Statistical Analysis 11: Comparison: Per-protocol Population; Family monthly income per capita, 5000 to 7999 RMB vs >=10000 RMB; Test type: Superiority or Other; p = 0.364, Chi-squared; Degrees of freedom=1, Wald Chi-Square=0.824; Odds Ratio (OR) = 1.060, 95% CI 2-sided [0.344 to 3.267]
Statistical Analysis 12: Comparison: Per-protocol Population; Test type: Superiority or Other; p = 0.175, Chi-squared; Degrees of freedom=1, Wald Chi-Square=1.838; Odds Ratio (OR) = 0.580, 95% CI 2-sided [0.100 to 3.347]
Statistical Analysis 13: Comparison: Per-protocol Population; Whether have brothers or sisters, no vs yes; Test type: Superiority or Other; p < 0.001, Chi-squared; Degrees of freedom=1, Wald Chi-Square=25.960; Odds Ratio (OR) = 0.516, 95% CI 2-sided [0.400 to 0.666]

9. Secondary Outcome: Risk Factors Associated With Nasopharyngeal Carriage for Haemophilus Influenzae Type B
Description: Risk factors include birth information (preterm vs full-term birth); household register (local vs nonlocal); feeding manners within 6 months (pure breast feeding, mixed feeding vs pure formula milk feeding); father's education level (illiteracy, elementary school, junior middle school, senior/vocational high school or technical, college/university vs postgraduate and above); living space per capita (continuous variables); vaccination history of Haemophilus influenzae type B (Hib) (no vs yes).
Time Frame: Day 1
Population: PP
Measure: Mean (Standard Error); unit: relative risk
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 3600
relative risk
  Birth information, preterm vs full-term birth | -0.683 (0.359)
  Household register, local vs nonlocal | -0.204 (0.099)
  Feeding, pure breast feeding vs pure formula milk | 0.227 (0.113)
  Feeding, mixed feeding vs pure formula milk | -0.287 (0.138)
  Father's education, illiteracy vs postgraduate | 2.857 (1.047)
  Father's education, elementary vs postgraduate | -0.126 (0.448)
  Father's education, junior middle vs postgraduate | -0.093 (0.298)
  Father's education, senior high vs postgraduate | -0.411 (0.306)
  Father's education, college vs postgraduate | -0.559 (0.316)
  Living space per capita, continuous variables | -0.016 (0.009)
  Vaccination history of Hib, no vs yes | -0.158 (0.085)
Statistical Analysis 1: Comparison: Per-protocol Population; Birth information, preterm birth vs full-term birth; Test type: Superiority or Other; p = 0.057, Chi-squared; Degrees of freedom=1, Wald Chi-Square=3.610; Odds Ratio (OR) = 0.255, 95% CI 2-sided [0.062 to 1.044]
Statistical Analysis 2: Comparison: Per-protocol Population; Household register, local vs nonlocal; Test type: Superiority or Other; p = 0.040, Chi-squared; Degrees of freedom=1, Wald Chi-Square=4.228; Odds Ratio (OR) = 0.666, 95% CI 2-sided [0.451 to 0.981]
Statistical Analysis 3: Comparison: Per-protocol Population; Feeding manners within 6 months, pure breast feeding vs pure formula milk feeding; Test type: Superiority or Other; p = 0.044, Chi-squared; Degrees of freedom=1, Wald Chi-Square=4.074; Odds Ratio (OR) = 1.182, 95% CI 2-sided [0.758 to 1.844]
Statistical Analysis 4: Comparison: Per-protocol Population; Feeding manners within 6 months, mixed feeding vs pure formula milk feeding; Test type: Superiority or Other; p = 0.038, Chi-squared; Degrees of freedom=1, Wald Chi-Square=4.316; Odds Ratio (OR) = 0.707, 95% CI 2-sided [0.420 to 1.191]
Statistical Analysis 5: Comparison: Per-protocol Population; Father's education level, illiteracy vs postgraduate or above; Test type: Superiority or Other; p = 0.006, Chi-squared; Degrees of freedom=1, Wald Chi-Square=7.438; Odds Ratio (OR) = 92.229, 95% CI 2-sided [3.993 to 2130.500]
Statistical Analysis 6: Comparison: Per-protocol Population; Father's education level, elementary school vs postgraduate or above; Test type: Superiority or Other; p = 0.778, Chi-squared; Degrees of freedom=1, Wald Chi-Square=0.079; Odds Ratio (OR) = 4.671, 95% CI 2-sided [0.537 to 40.608]
Statistical Analysis 7: Comparison: Per-protocol Population; Father's education level, junior high school vs postgraduate or above; Test type: Superiority or Other; p = 0.756, Chi-squared; Degrees of freedom=1, Wald Chi-Square=0.096; Odds Ratio (OR) = 4.830, 95% CI 2-sided [0.649 to 35.956]
Statistical Analysis 8: Comparison: Per-protocol Population; Father's education level, senior high school/vocational high school/technical secondary school vs postgraduate or above; Test type: Superiority or Other; p = 0.179, Chi-squared; Degrees of freedom=1, Wald Chi-Square=1.807; Odds Ratio (OR) = 3.513, 95% CI 2-sided [0.474 to 26.030]
Statistical Analysis 9: Comparison: Per-protocol Population; Father's education level, college/university vs postgraduate or above; Test type: Superiority or Other; p = 0.077, Chi-squared; Degrees of freedom=1, Wald Chi-Square=3.131; Odds Ratio (OR) = 3.029, 95% CI 2-sided [0.412 to 22.292]
Statistical Analysis 10: Comparison: Per-protocol Population; Living space per capita, continuous variables; Test type: Superiority or Other; p = 0.056, Chi-squared; Degrees of freedom=1, Wald Chi-Square=3.648; Odds Ratio (OR) = 0.984, 95% CI 2-sided [0.968 to 1.000]
Statistical Analysis 11: Comparison: Per-protocol Population; Vaccination history of Hib, no vs yes; Test type: Superiority or Other; p = 0.064, Chi-squared; Degrees of freedom=1, Wald Chi-Square=3.432; Odds Ratio (OR) = 0.729, 95% CI 2-sided [0.522 to 1.018]

10. Secondary Outcome: Risk Factors Associated With Nasopharyngeal Carriage for Moraxella Catarrhalis
Description: Risk factors include birth information (preterm vs full-term birth); household register (local vs nonlocal); mother's education level (illiteracy, elementary school, junior middle school, senior/vocational high school or technical, college/university, vs postgraduate and above); whether have brothers or sisters (no vs yes).
Time Frame: Day 1
Population: PP
Measure: Mean (Standard Error); unit: relative risk
Arm/Group | Per-protocol Population
Number analyzed (Participants) | 3600
relative risk
  Birth information, preterm vs full-term birth | -0.412 (0.175)
  Household register, local vs nonlocal | -0.303 (0.065)
  Mother's education, illiteracy vs graduate | 0.280 (0.479)
  Mother's education, elementary vs graduate | 0.104 (0.214)
  Mother's education, junior middle vs graduate | 0.199 (0.153)
  Mother's education, senior high vs postgraduate | 0.166 (0.159)
  Mother's education, college vs postgraduate | -0.270 (0.174)
  Whether have brothers or sisters, no vs yes | -0.203 (0.063)
Statistical Analysis 1: Comparison: Per-protocol Population; Birth information, preterm birth vs full-term birth; Test type: Superiority or Other; p = 0.019, Chi-squared; Degrees of freedom=1, Wald Chi-Square=5.538; Odds Ratio (OR) = 0.438, 95% CI 2-sided [0.221 to 0.871]
Statistical Analysis 2: Comparison: Per-protocol Population; Household register, local vs nonlocal; Test type: Superiority or Other; p < 0.001, Chi-squared; Degrees of freedom=1, Wald Chi-Square=21.938; Odds Ratio (OR) = 0.546, 95% CI 2-sided [0.423 to 0.703]
Statistical Analysis 3: Comparison: Per-protocol Population; Mother's education level, illiteracy vs graduate or above; Test type: Superiority or Other; p = 0.559, Chi-squared; Degrees of freedom=1, Wald Chi-Square=0.341; Odds Ratio (OR) = 2.137, 95% CI 2-sided [0.473 to 9.652]
Statistical Analysis 4: Comparison: Per-protocol Population; Mother's education level, elementary school vs graduate or above; Test type: Superiority or Other; p = 0.626, Chi-squared; Degrees of freedom=1, Wald Chi-Square=0.238; Odds Ratio (OR) = 1.793, 95% CI 2-sided [0.596 to 5.394]
Statistical Analysis 5: Comparison: Per-protocol Population; Mother's education level, junior middle school vs graduate or above; Test type: Superiority or Other; p = 0.193, Chi-squared; Degrees of freedom=1, Wald Chi-Square=1.691; Odds Ratio (OR) = 1.972, 95% CI 2-sided [0.699 to 5.562]
Statistical Analysis 6: Comparison: Per-protocol Population; Mother's education level, senior high school/vocational high school/technical secondary school vs postgraduate or above; Test type: Superiority or Other; p = 0.298, Chi-squared; Degrees of freedom=1, Wald Chi-Square=1.081; Odds Ratio (OR) = 1.907, 95% CI 2-sided [0.679 to 5.353]
Statistical Analysis 7: Comparison: Per-protocol Population; Mother's education level, college/university vs postgraduate or above; Test type: Superiority or Other; p = 0.122, Chi-squared; Degrees of freedom=1, Wald Chi-Square=2.395; Odds Ratio (OR) = 1.233, 95% CI 2-sided [0.439 to 3.464]
Statistical Analysis 8: Comparison: Per-protocol Population; Whether have brothers or sisters, no vs yes; Test type: Superiority or Other; p = 0.001, Chi-squared; Degrees of freedom=1, Wald Chi-Square=10.233; Odds Ratio (OR) = 0.666, 95% CI 2-sided [0.520 to 0.855]

ADVERSE EVENTS:
Arm/Group | Per-protocol Population
Serious Adverse Events (participants affected / at risk) | 0/3600
Other Adverse Events (participants affected / at risk) | 0/3600

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wyeth has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.